CLINICAL TRIAL: NCT06190990
Title: Additional Effects of Otago Exercises With Exer-gaming on Balance, Physical Performance and Gait Among the Elderly Population
Brief Title: Otago Exercises and Otago Exercise Effects on Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jalwa Zahid
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Elderly Population
Keywords: Exer gaming; Otago exercises; Distorted balance; Disturbed gait; Reduce physical performance; Older population

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- additional effects of exer gaming with otago exercises (Other): Strengthening training
  * Sitting knee extension
  * Standing hip abduction
  * Standing knee flexion
  * Tip toe
  * Heel tiptoe Balance training
  * Knee bends
  * Backward walking
  * Walk in figure 8
  * Sideways walking
  * Tandem stands
  * Tandem walking
  * 1-leg stand
  * Heel walking
  * Toe walking
  * Heel-toe walking backward
  * Sit to stand After Otago exercises, the participants will receive the following exer-gaming based exercises.
  * Football player
  * Boat
  * Volleyball beach
  Interventions: Other: Otago Exercise + Exer gaming
- exer gaming based exercises (Other): The participants will receive the following exer-gaming based exercises.
  * Football player
  * Boat
  * Volleyball beach
  Interventions: Other: exer gaming based programme

INTERVENTIONS:
Other: Otago Exercise + Exer gaming — In this group the participant will receive otago exercises and exer-gaming based exercises. The duration of each session this group will receive is of 60 minutes A total of 12 sessions will be held, 3 times a week for 4 weeks. Reading will be taken on baseline, after 2 week
  Arms: additional effects of exer gaming with otago exercises
Other: exer gaming based programme — In this group the participant will receive exer-gaming based exercises. The duration of each session this group will receive is of 60 minutes A total of 12 sessions will be held, 3 times a week for 4 weeks. Reading will be taken on baseline, after 2 weeks and then after 4 weeks.
  Arms: exer gaming based exercises

SUMMARY:
Study aims to investigate the profound impact of exer gaming on normal aged individuals within our society. Additionally, to compare the effects of exer gaming-based exercises and Otago exercises on crucial aspects such as balance, physical performance, and gait pattern among the normal aged population. This study holds immense significance as it has the potential to greatly improve the health and wellbeing of the elderly population. By identifying an efficacious physical therapy intervention to address the complications associated with balance, physical performance, and gait pattern, we can effectively mitigate further dysfunctions in this demographic.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age > 55 Years
* Berg balance scale score 21-40
* Moca >24
* Urinary bowel continence

Exclusion Criteria:

* Having history of other neurological conditions (i.e. Dementia, Parkinson's disease)
* Having contagious or inflammatory conditions.
* Having orthopedic limitations such as fractures
* Unable to comply with the training or currently participating in another interfering therapy
* With Vision problems
* Having uncontrolled cardiac conditions such as uncontrolled hypertension

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 4th week
  Consists of 14 tasks and total score of 56.score of 0-20 indicates severe fall risk, 20-45 includes moderate risk of fall and 45-60 illustrates thr functional balances state.

SECONDARY OUTCOMES:
Time Up and Go (TUG) | 4th week
  The TUG test is a simple assessment used to evaluate a person's mobility and balance. It measures the time it takes for an individual to stand up from a seated position, walk a short distance (typically 3 meters), turn around, walk back, and sit down again. This test is often used to assess the risk of falls among older adults
dynamic gait index | 4th week
  Assess the likelihood of falling in older adults.total score is of 24.score less than 19 is predictive of fall risks.
10 Meter Walk Test (10MWT) | 4th week
  The 10MWT is a clinical assessment used to measure an individual's walking speed over a 10-meter distance. It is often used to assess gait and mobility, as well as to track changes in a person's walking abilities over time.
Montreal Cognitive Assessment | 4th week
  Montreal Cognitive Assessment (MoCA) is a cognitive assessment tool used to screen for mild cognitive impairment. It assesses various cognitive functions, including memory, attention, language, and visuospatial abilities. It consists of tasks and questions that provide a total score, with lower scores indicating potential cognitive deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- RAFSAN Neuro Rehabilitation center, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No